CLINICAL TRIAL: NCT02817971
Title: Effect of Enhanced Feedback to Hospitals That Are Part of an Emerging Clinical Information Network on Uptake of Revised Childhood Pneumonia Treatment Policy: A Pragmatic Cluster Randomized Trial Protocol
Brief Title: Effect of Enhanced Feedback to Hospitals in an Emerging Clinical Information Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KEMRI_CT_2016\0021
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Pneumonia
Keywords: feedback; pneumonia; quality of care
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced feedback (Experimental): 1. Monthly written feedback incorporating goal setting, and action planning delivered by a senior clinical coordinator for selected pneumonia indicators
  2. Two-monthly written feedback on multiple quality of paediatric care indicators
  3. Clinical network promoting clinical leadership linked to mentorship and peer to peer support
  4. Improved use of health information on service delivery
  Interventions: Behavioral: Enhanced feedback
- Standard feedback (Active Comparator): 1. Two-monthly written feedback on multiple quality of paediatric care indicators
  2. Clinical network promoting clinical leadership linked to mentorship and peer to peer support
  3. Improved use of health information on service delivery
  Interventions: Behavioral: Standard feedback

INTERVENTIONS:
Behavioral: Enhanced feedback — Hospital level feedback delivered every month through paediatrician on the level of adherence to revised pneumonia treatment recommendations.
  Arms: Enhanced feedback
Behavioral: Standard feedback — Hospital level feedback delivered every two months through paediatrician on the performance of multiple paediatric care indicators for managing severely ill children.
  Arms: Standard feedback

SUMMARY:
A cluster randomised pragmatic trial will be conducted within an emerging clinical information network composed of 12 Kenyan county hospitals. Hospitals will be randomised to an enhanced feedback intervention delivered over a nine-month period and compared to standard feedback. The trial to be implemented during a phase of implementing change in guideline recommendations for pneumonia will assess the impact of enhanced feedback on hospital uptake of the revised pneumonia treatment recommendations.

DETAILED DESCRIPTION:
The international guidelines for the classification and treatment of childhood pneumonia were revised recently and in Kenya the national guidelines changed in February 2016. We designed an enhanced feedback intervention aimed at improving uptake of the revised pneumonia treatment policy within a clinical network of 12 Kenyan county referral hospitals.

Hospitals were randomized to receive either enhanced feedback (n = 6 hospitals) or standard feedback (n = 6 hospitals) delivered over a six-month period following nationwide pneumonia treatment policy change. The primary outcome is the proportion of all pneumonia admissions (fulfilling criteria for treatment with oral amoxicillin) who are correctly classified and treated using new guideline recommendations. The proportion of treatment change from oral amoxicillin to alternative antibiotics for pneumonia (considered a proxy measure of treatment failure) will be reported as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 59 months admitted to participating network hospitals with WHO pneumonia diagnosis eligible for treatment with oral amoxicillin

Exclusion Criteria:

* Children aged 2 to 59 months with WHO pneumonia diagnosis and co-morbid illnesses requiring intravenous antibiotic treatment including severe acute malnutrition, bacteraemia, meningitis, or
* children presenting with pneumonia and tuberculosis or cough lasting more than 2 weeks, or severe malaria

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pneumonia classification and treatment | 9 months
  The proportion of all pneumonia admissions (fulfilling criteria for treatment with oral amoxicillin) who are correctly classified and treated using new guideline recommendations

SECONDARY OUTCOMES:
Antibiotic change | 9 months
  The proportion of treatment change from oral amoxicillin to alternative antibiotics for pneumonia (considered a proxy measure of treatment failure)

CONTACTS AND LOCATIONS:
Overall Officials: Mike English, MD, Principal Investigator — KEMRI-Wellcome Trust Research Priogramme
Locations (12):
- Kenya (12):
  - Kerugoya County Hospital, Kerugoya, Kerugoya
  - Busia County Hospital, Busia
  - Embu County Hospital, Embu
  - Kakamega County Referral Hospital, Kakamega
  - Vihiga County Hospital, Kakamega
  - Karatina County Hospital, Karatina
  - Kiambu County Hospital, Kiambu
  - Kisumu County Hospital, Kisumu
  - Kitale County Hospital, Kitale
  - Machakos County Hospital, Machakos
  - Mama Lucy Kibaki Hospital, Nairobi
  - Nyeri County Hospital, Nyeri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayieko P, Irimu G, Ogero M, Mwaniki P, Malla L, Julius T, Chepkirui M, Mbevi G, Oliwa J, Agweyu A, Akech S, Were F, English M; Clinical Information Network Authors. Effect of enhancing audit and feedback on uptake of childhood pneumonia treatment policy in hospitals that are part of a clinical network: a cluster randomized trial. Implement Sci. 2019 Mar 4;14(1):20. doi: 10.1186/s13012-019-0868-4. PMID 30832678
- [Derived] Ayieko P, Irimu G, English M. Effect of enhanced feedback to hospitals that are part of an emerging clinical information network on uptake of revised childhood pneumonia treatment policy: study protocol for a cluster randomized trial. Trials. 2017 Sep 7;18(1):416. doi: 10.1186/s13063-017-2152-8. PMID 28877729